CLINICAL TRIAL: NCT02514889
Title: Is MyPlate.Gov Approach to Helping Overweight Patients Lose Weight More Patient-centered?
Brief Title: Is MyPlate Approach to Helping Overweight Patients Lose Weight More Patient-centered?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, William J. McCarthy, Ph.D., Adjunct Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PCORI-1306-01150
Record Dates: First submitted 2015-04-18; First posted 2015-08-04 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calorie-counting (Active Comparator): Intervention protocol adapted from Diabetes Prevention Program lifestyle change intervention.
  Interventions: Behavioral: Calorie-counting
- MyPlate (Experimental): Intervention protocol adapted from Dietary Approaches to Stop Hypertension dietary pattern.
  Interventions: Behavioral: MyPlate

INTERVENTIONS:
Behavioral: Calorie-counting — The Calorie Counting (CC) condition asks obese patients to achieve a daily calorie deficit. For average women consuming 2,000 calories at baseline, the target daily calorie total might be 1,600 calories. Participants are also asked to do at least 150 minutes of moderate to vigorous physical activity per week.
  Two community health workers will provide behavior change coaching to 150 TCC obese patients randomly assigned to the CC condition. The intervention protocol is adapted from the Diabetes Prevention Program. Behavior change strategies include: self-monitoring (e.g., calorie-counting, self-weighing), stimulus control, and relapse prevention strategies. The health coaching will occur during two home visits, two group health education sessions, and 7 telephone coaching calls.
  Other Names: DPP intensive lifestyle change intervention
  Arms: Calorie-counting
Behavioral: MyPlate — The MyPlate approach asks Americans to limit daily calories but emphasizes eating MORE high-satiation foods by making ½ of daily food choices fruits and vegetables,¼ of daily food choices whole grains. All participants are asked to do at least 150 minutes of moderate to vigorous physical activity per week.
  Two community health workers will provide behavior change coaching to 150 TCC obese patients randomly assigned to the MyPlate condition. MyPlate is adapted from the DASH protocol. Behavior change strategies include: progressive goal-setting, stimulus control, and self-monitoring (e.g., % of food choices that are fruits & vegetables). The health coaching will occur during two home visits, two group health education sessions, and 7 telephone behavior change coaching calls.
  Other Names: DASH diet intervention
  Arms: MyPlate

SUMMARY:
Investigators from the University of California-Los Angeles (UCLA) and The Children's Clinic of Long Beach (TCC) are conducting a randomized, controlled comparative effectiveness trial of two government-sanctioned behavior change approaches to weight control with TCC's obese patients. The first approach is the calorie-counting calorie restriction (CC) approach used in the Diabetes Prevention Program. The second approach is the high-satiation/high-satiety approach represented by MyPlate.gov. The MyPlate nutritional goal is to double patient fruit and vegetable intake, legume intake, and whole grain intake. Both conditions stipulate 150 minutes of moderate physical activity a week. Study participants will be 300 of TCC's obese patients, 76% of whom are expected to be Latino, 13% African American and 11% Other Ethnicities.

The interventions will be implemented by trained community lifestyle change coaches with brief support from clinicians. The interventions will include two home visits, two group education sessions and seven telephone behavior change coaching sessions.

Compared to the CC approach, the MyPlate approach is hypothesized to yield better 12 months patient-centered outcomes, particularly self-reported satiety.

DETAILED DESCRIPTION:
The traditional government advice for weight loss in obese patients has been calorie-counting(CC) / portion control. In 2011 the government began recommending the MyPlate approach (MyP) for optimal nutrition and better weight control. The CC condition asks obese patients to reduce their daily calorie intake to less than a recommended calorie target. The MyP approach also limits daily calories but emphasizes eating MORE high-satiation foods by making ½ of daily food choices fruits and vegetables, and ¼ of daily food choices whole grains. The relative patient-centered outcome effectiveness of the MyP approach versus the CC approach has yet to be tested in clinic patients.

Specific Aims:

In partnership with a local community clinic, the investigators are conducting a randomized controlled trial (RCT) comparing the patient-centeredness and efficacy of usual care compared to two government-supported lifestyle change approaches to reducing patient obesity risk. Study participants are 300 obese, low income, mostly Latino and African American adult patients or staff associated with a community health center in Long Beach, California. The interventions will be implemented by trained community lifestyle change coaches with brief support from clinicians.

The first weight loss approach is the calorie-counting (CC), portion-cutting approach recommended at www.nutrition.gov . The second is the fill-up-sooner-on-fewer-calories approach found at http://www.choosemyplate.gov (MyP). The CC condition asks overweight patients to reduce their daily calorie intake to less than a recommended calorie target. The MyP approach also limits daily calories but emphasizes eating MORE high-satiation foods by making ½ of daily food choices fruits and vegetables, and ¼ of daily food choices whole grains. MyP uses progressive goal-setting to facilitate a doubling of usual fruit and vegetable intake. To facilitate adherence, the MyP approach also includes home environment changes to make healthier choices easier choices. All conditions encourage doing at least 150 minutes of moderate to vigorous physical activity a week. Primary patient-centered outcomes include self-reported satiety, health-related quality of life, self-efficacy to eat more fruits and vegetables, patient autonomy, and patient satisfaction, all of which are hypothesized to favor the MyP condition at 12 months follow-up relative to the CC condition. The primary medical outcome is a reduction in body weight.

Specific Aims Aim #1. Use qualitative information from patients and clinical staff to revise intervention materials and procedures. Aim #2. Use results of a pilot test of the intervention conditions to revise intervention materials and procedures. Aim #3. Conduct a 1-year RCT involving two home visits, two group education classes, and seven telephone support/ lifestyle change coaching calls. Aim #4. Obtain qualitative data from providers and coaches; combine with participant data to assess intervention feasibility, acceptability and perceived usefulness. Aim #5. Disseminate results and recommendations to community groups and public health professionals.

Primary patient-centered hypothesis: Compared to the CC approach, the MyP approach will yield better 1-year outcomes on self-reported satiety and systolic blood pressure. Both government-recommended conditions will yield significant and similar 12 months declines in body weight.

The MyPlate distillation of the 2010 Dietary Guidelines for Americans shifted the emphasis of nutrition recommendations for desirable weight loss from counting calories to maximizing satiation, through the practical steps of eating MORE fruits and vegetables, MORE whole grains, MORE nonfat dairy, MORE water (and LESS sugary beverages). Calorie counting helps lose excess weight in the short term but rarely is able to sustain desirable weight loss long-term. The MyPlate approach may be easier to sustain because it allows eating up to 25 percent more grams of food even as it reduces baseline calorie intake by 10 percent; the extra daily grams of food help the patient to feel full even while she is losing weight. Because MyPlate is a distillation of recommendations for all healthy Americans, regardless of body size, it can guide eating choices for everyone in the family and do so for a lifetime. If the MyPlate approach is shown to be as effective in helping patients to sustain 1-year weight loss as the DPP approach, more clinicians can be expected to actively engage their obese patients in weight loss efforts.

ELIGIBILITY:
Inclusion Criteria:

* Must be overweight (BMI > 25) or obese adult patient at The Childrens Clinic of Long Beach (TCC),
* interested in achieving desirable weight loss through behavior change.
* speak English or Spanish.

Exclusion Criteria:

* Smoking in last 6 months,
* Currently pregnant,
* Medical condition preventing voluntary change in food choices or level of daily physical activity,
* Planning on moving out of the Long Beach area in the next two years.
* MyocardiaI Infarction, stroke or atherosclerotic cardiovascular disease procedure within the last 6 months
* Serious medical condition likely to hinder accurate measurement of weight, or for which weight loss is contraindicated, or which would cause weight loss (e.g. End Stage Renal Disease on dialysis, cancer diagnosis or treatment within 2 yrs)
* Prior or planned bariatric surgery
* Use of prescription weight loss medication (including off label drugs e.g. topiramate, bupropion, byetta) or over-the-counter orlistat within 6 months
* Chronic use (at least past 6 months) of medications likely to cause weight gain or prevent weight loss (e.g. corticosteroids, lithium, olanzapine, risperidone, clozapine)
* Unintentional weight loss within past 6 months (≥ 5% of body weight)
* Intentional weight loss within past 6 months (≥ 5% of body weight)
* Pregnant or nursing within past 6 months
* Plans to become pregnant within 18 months
* Another member of household is a study participant or trial staff member
* Problem alcohol use: Self reported average consumption of > 14 alcoholic drink per week or 5+ drinks on any occasion in past week? for males and >7 drinks per week or 4+ drinks on any occasion in the past week for females
* Psychiatric hospitalization in last year
* Unstable angina
* Blood pressure >160/100 (note: individuals may be rescreened)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J McCarthy, Ph.D., Principal Investigator — UCLA Fielding School of Public Health
Locations (2):
- United States (2):
  - The Children's Clinic of Long Beach (TCC), Long Beach, California
  - UCLA Center for Cancer Prevention & Control Research, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Yes
The Fielding School of Public Health Open Data Portal is a web application being built that will enable the sharing of public health research, data and data tools. The platform operates in a secure, HIPPA compliant, cloud environment. The project's de-identified data, protocol and codebook will remain stored in an encrypted form. The portal was expressly designed to make new public health data available through a creative commons framework, available to any researcher willing to comply with UCLA IRB stipulations.
Supporting Information: Study Protocol, ICF
Time Frame: By 6/30/2018.
Access Criteria: UCLA IRB approval required.

REFERENCES:
- [Derived] Gelberg L, Rico MW, Herman DR, Belin TR, Chandler M, Ramirez E, Love S, McCarthy WJ. Comparative effectiveness trial comparing MyPlate to calorie counting for mostly low-income Latino primary care patients of a federally qualified community health center: study design, baseline characteristics. BMC Public Health. 2019 Jul 24;19(1):990. doi: 10.1186/s12889-019-7294-z. PMID 31340800

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All adult patients in waiting room of two clinics were approached for assessment of eligibility to enroll in the trial. The eligibility assessment period began 4/1/2015 and ended on 2/5/2016. 2,086 patients were approached; screening was completed for 1,889. Of these 1,889, 1,628 were found to be ineligible, leaving 261 to be randomized.
Pre-assignment Details: All participants who were enrolled were randomized.
Groups:
- MyPlate: Intervention protocol adapted from Dietary Approaches to Stop Hypertension dietary pattern.
  MyPlate: The MyPlate approach asks Americans to limit daily calories but emphasizes eating MORE high-satiation foods by making ½ of daily food choices fruits and vegetables,¼ of daily food choices whole grains. All participants are asked to do at least 150 minutes of moderate to vigorous physical activity per week.
  Two community health workers will provide behavior change coaching to 150 TCC obese patients randomly assigned to the MyPlate condition. MyPlate is adapted from the DASH protocol. Behavior change strategies include: progressive goal-setting, stimulus control, and self-monitoring (e.g., % of food choices that are fruits & vegetables). The health coaching will occur during two home visits, two group health education sessions, and 7 telephone behavior change coaching calls.
- Calorie-counting: Intervention protocol adapted from Diabetes Prevention Program lifestyle change intervention.
  Calorie-counting: The Calorie Counting (CC) condition asks obese patients to achieve a daily calorie deficit. For average women consuming 2,000 calories at baseline, the target daily calorie total might be 1,600 calories. Participants are also asked to do at least 150 minutes of moderate to vigorous physical activity per week.
  Two community health workers will provide behavior change coaching to 150 TCC obese patients randomly assigned to the CC condition. The intervention protocol is adapted from the Diabetes Prevention Program. Behavior change strategies include: self-monitoring (e.g., calorie-counting, self-weighing), stimulus control, and relapse prevention strategies. The health coaching will occur during two home visits, two group health education sessions, and 7 telephone coaching calls.
Period: Randomization/Allocation to Condition
Arm/Group | MyPlate | Calorie-counting
Started | 131 | 130
Completed | 111 | 106
Not Completed | 20 | 24
Period: Intervention Participation
Arm/Group | MyPlate | Calorie-counting
Started | 111 | 106
Completed | 102 | 98
Not Completed | 9 | 8
Period: Follow-up Assessment Participation
Arm/Group | MyPlate | Calorie-counting
Started (179 participants provided survey data via in-person interviews; 21 provided survey data via phone) | 102 | 98
Completed (179 participants completed in-person follow-up but 1 in-person visit did not include waist measure) | 92 | 86
Not Completed | 10 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MyPlate | Calorie-counting | Total
Number analyzed (Participants) | 131 | 130 | 261
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (11.5) | 41.8 (11.5) | 41.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 123 | 249
  Male | 5 | 7 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: African American | 10 | 10 | 20
  Ethnicity: Asian American | 1 | 1 | 2
  Ethnicity: Non-Hispanic White | 7 | 3 | 10
  Ethnicity: Hispanic/Latino | 112 | 113 | 225
  Ethnicity: Native American | 0 | 1 | 1
  Ethnicity: Other | 1 | 2 | 3
Region of Enrollment [Number; unit: Count of participants]
  United States | 131 | 130 | 261
Hunger level yesterday [Mean (Standard Deviation); unit: Units on a scale] — Primary patient-centered outcome measure was response to question: "Thinking about yesterday, how hungry did you feel during the day?" Response was a mark on a 100mm scale, 0="Not at all hungry" and 100="Extremely hungry."
  Units on a scale | 47.11 (27.46) | 51.01 (27.36) | 49.05 (27.43)
Meal satisfaction yesterday [Mean (Standard Deviation); unit: Units on a scale] — Response to question "Take a moment to think about the last meal you ate yesterday. Thinking about the last meal you ate, how satisfied were you after you ate that meal?", marked on a 100 mm visual analogue scale, with 0="Very satisfied" 100="Very unsatisfied anchoring the high end of the scale, and reverse-coded for analysis, so that higher values (up to 100) represent greater meal satisfaction than lower values (as low as 0).
  Units on a scale | 66.69 (2.88) | 69.15 (2.88) | 67.92 (2.03)
Feeling full after last meal yesterday [Mean (Standard Deviation); unit: units on a scale] — Response to the question "Take a moment to remember the last meal you ate yesterday. Thinking about the last meal you ate, how full did you feel after you ate that meal?" Response was recorded on a 100mm visual analogue scale, with "Extremely full" anchoring the low end of the scale (0) and "Not at all full" anchoring the high end of the scale (100). For analysis purposes this measure was reverse-scored, so that greater values represent greater fullness ratings.
  units on a scale | 66.05 (29.34) | 69.92 (28.50) | 67.97 (28.93)
Body weight (kg) [Mean (Standard Deviation); unit: kg] | 81.17 (0.95) | 83.29 (0.72) | 82.23 (0.72)
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 32.98 (0.32) | 33.66 (0.32) | 33.32 (0.23)
Waist circumference (cm) [Mean (Standard Deviation); unit: cm] — The waist circumference measure was variably taken against the skin and taken over clothing, depending on patient preference. On average, collecting waist circumference over clothing appeared to add 3.47cm to measurements. The measure reported here does not correct for this error but measures that did subtract 3.47 cm from all waist circumference measurements taken over light clothing did not yield different findings compared to the findings based on uncorrected waist circumference measures. Population: At beginning of study one female patient refused to have her waist circumference taken by the only research assistant available at the time, who was male, which resulted in loss of data. We subsequently permitted the taking of waist circumference measures over clothing depending on patient preference.
  cm
    number analyzed (Participants) | 130 | 130 | 260
    (all) | 100.60 (0.78) | 103.47 (0.85) | 102.03 (0.58)
Systolic blood pressure [Mean (Standard Deviation); unit: mm (mercury-equivalent)] | 122.19 (1.24) | 122.67 (1.40) | 122.43 (0.93)

OUTCOME MEASURES:

1. Primary Outcome: Patient-centered Outcome Measure = Self-reported Hunger
Description: Response to question: "Thinking about yesterday, how hungry did you feel during the day?" Response was a mark on a 100mm scale or oral response on a scale from 0 to 100 (for participants assessed via phone), 0="Not at all hungry" and 100="Extremely hungry."
Time Frame: 12 months follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MyPlate | Calorie-counting
Number analyzed (Participants) | 102 | 98
units on a scale | 40.6 (2.33) | 40.8 (2.14)
Statistical Analysis 1: Comparison: MyPlate vs Calorie-counting; Test type: Superiority; p = 0.30, Mixed Models Analysis — a priori threshold is p = .017, so that experiment-wide critical alpha would be p = .05; Covariates: sex, age, ethnicity, marital status and educational attainment; Mean Difference (Final Values) = -2.11, 95% CI 2-sided [-6.12 to 1.91], Standard Error of Mean 2.05 — Difference in differences interaction term is the product of assessment period (baseline, 6-months, 12-months) and experimental condition (MyPlate, Calorie Counting)

2. Primary Outcome: Medical Outcome Measure = Body Weight
Description: Body weight, measured in kilograms, was obtained by having shoeless participants dressed in light clothing stand on a regularly calibrated medical scale. Measures were taken twice. If these measures differed by more than 0.2 kg, a third measure was taken and averaged with the other two.
Time Frame: 12 months follow-up
Population: Participants who completed the in-person follow-up visit for anthropometric evaluation
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | MyPlate | Calorie-counting
Number analyzed (Participants) | 93 | 86
kilograms | 80.5 (1.19) | 82.6 (1.48)
Statistical Analysis 1: Comparison: MyPlate vs Calorie-counting; Test type: Equivalence — p-value >0.20 would be considered equivalent; p = 0.06, Mixed Models Analysis; Covariates included age, sex, ethnicity, educational attainment and marital status; Mean Difference (Final Values) = 2.59, 95% CI 2-sided [-0.1342 to 5.3228], Standard Error of Mean 1.39

3. Primary Outcome: Meal Satisfaction Yesterday
Description: "Take a moment to think about the last meal you ate yesterday. Thinking about the last meal you ate, how satisfied were you after the meal?" Response was a mark on a 100 mm visual analogue scale or response to oral question on a scale from 0 to 100 (for participants assessed via phone), with the low end (0) anchored by "Very satisfied" and the high end (100) anchored by "Very unsatisfied." For analysis purposes this measure was reverse-scored, so that higher values represented greater meal satisfaction.
Time Frame: 12 months follow-up
Population: Participants who provided survey data at follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MyPlate | Calorie-counting
Number analyzed (Participants) | 102 | 98
units on a scale | 83.4 (2.51) | 83.5 (2.48)
Statistical Analysis 1: Comparison: MyPlate vs Calorie-counting; Test type: Superiority; p = 0.504, Mixed Models Analysis; Covariates included: age, sex, ethnicity, educational attainment and marital status; Mean Difference (Net) = -1.37, 95% CI 2-sided [-6.37 to 3.63], Standard Error of Mean 2.55 — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Feeling Full After Last Meal Yesterday
Description: "Take a moment to think about the last meal yesterday. Thinking about the last meal you ate, how full did you feel after that meal?" Response was a mark on a 100 mm visual analogue scale (VAS), or oral response to question on a scale from 0 to 100 (for participants assessed via phone), 0="Extremely full" and 100="Not at all full." For analysis purposes this measure was reverse-scored, so that higher values represented greater fullness.
Time Frame: 12 months follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MyPlate | Calorie-counting
Number analyzed (Participants) | 102 | 98
units on a scale | 78.6 (2.10) | 78.6 (2.51)
Statistical Analysis 1: Comparison: MyPlate vs Calorie-counting; Test type: Superiority — Difference in differences; p = 0.30, Mixed Models Analysis; Covariates included: age, sex, ethnicity, educational attainment, marital status; Mean Difference (Net) = -1.88, 95% CI 2-sided [-6.47 to 2.74], Standard Error of Mean 2.35 — The difference in differences interaction term is the product of assessment period (baseline, 6-months, 12-months) and experimental condition (MyPlate, Calorie Counting)

5. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure assessed on participant's left arm while participant is seated, after at least 5 minutes of rest. Automated, regularly calibrated sphygmomanometer was used with oversize cuffs for obese arms.
Time Frame: 12 months follow-up
Population: Participants who completed in-person evaluation at 12 months follow-up
Measure: Mean (Standard Error); unit: mm of mercury (equivalent)
Arm/Group | MyPlate | Calorie-counting
Number analyzed (Participants) | 93 | 86
mm of mercury (equivalent) | 121.6 (1.43) | 123.4 (2.05)
Statistical Analysis 1: Comparison: MyPlate vs Calorie-counting; Test type: Superiority; p = 0.640, Mixed Models Analysis; Mean Difference (Net) = 0.46, 95% CI 2-sided [-1.47 to 2.39], Standard Error of Mean 0.99 — The differences in difference interaction term consists of the product of assessment intervals (baseline, 6-months, 12-months) and experimental condition (MyPlate, Calorie Counting)

6. Secondary Outcome: Body Mass Index
Description: Body mass index is weight in kilograms divided by the square of the participant's height measured in meters. Wall-mounted stadiometer was used to assess height. Weekly-calibrated, portable, digital scales were used to assess body weight.
Time Frame: 12 months follow-up
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | MyPlate | Calorie-counting
Number analyzed (Participants) | 93 | 86
kg/m^2 | 33.25 (0.3457) | 34.01 (0.3496)
Statistical Analysis 1: Comparison: MyPlate vs Calorie-counting; Test type: Equivalence — For the comparison conditions to be equivalent, as predicted, the critical alpha was set at P > 0.20; p = 0.747, Mixed Models Analysis; Covariates included: age, sex, ethnicity, educational attainment and marital status; Mean Difference (Net) = -.04, 95% CI 2-sided [-.31 to 0.22], Standard Error of Mean 0.135 — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Waist Circumference
Description: The waist circumference was assessed using research standard waist circumference measuring tapes. The result was measured to closest 0.1 cm. The assessor was instructed to position the measuring tape horizontally around the waist, just above the iliac crest.
Time Frame: 12 months follow-up
Population: Of 93 participants completing in-person follow-up visit, 1 participant did not undergo waist measurement
Measure: Mean (Standard Error); unit: cm
Arm/Group | MyPlate | Calorie-counting
Number analyzed (Participants) | 92 | 86
cm | 98.6 (0.91) | 101.6 (1.12)
Statistical Analysis 1: Comparison: MyPlate vs Calorie-counting; Test type: Equivalence — For the comparison conditions to be judged equivalent, as predicted, the critical p-value was set to P >.20; p = 0.776, Mixed Models Analysis; Covariates included: age, sex, ethnicity, educational attainment and marital status; Mean Difference (Net) = 0.14, 95% CI 2-sided [-0.85 to 1.14], Standard Error of Mean 0.51 — [estimate comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: Participants were heavily monitored during the intervention phase, usually months 1-3 of their participation and then lightly for assessment-only purposes for months 4-12.
Description: Because the intervention evaluated federal lifestyle recommendations intended for application to all healthy adults, a data safety monitoring board was not established to oversee this particular trial. A health safety officer did agree to provide independent oversight of all adverse events associated with this trial.
Arm/Group | Calorie-counting | MyPlate
All-Cause Mortality (participants affected / at risk) | 0/130 | 1/131
Serious Adverse Events (participants affected / at risk) | 0/130 | 1/131
Other Adverse Events (participants affected / at risk) | 1/130 | 0/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calorie-counting (N=130) | MyPlate (N=131)
Death (General disorders) | 0 (0) | 1 (1) — Unconfirmed death reported by husband as reason why spouse was no longer participating. No cause of death was reported.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calorie-counting (N=130) | MyPlate (N=131)
Medical issues (unspecified) (General disorders) | 1 (1) | 0 (0) — Patient reported unspecified medical issues impeding her ability to continue participating in the trial. She made it clear that she did not consider these medical issues to have resulted from her participation in this study.

LIMITATIONS AND CAVEATS:
The original recruitment goal was N=300 but was reduced to N=261 because accrual took longer than expected. Statistical power was nonetheless expected to remain satisfactory for testing the main hypotheses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/89/NCT02514889/Prot_SAP_000.pdf
  • Informed Consent Form (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/89/NCT02514889/ICF_001.pdf